CLINICAL TRIAL: NCT05975268
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Subcutaneous JS005 Injection in the Treatment of Adults With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Subcutaneous JS005 Injection in the Treatment of Adults With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS005-005-III-PsO
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study uses a double-blind design in which subjects, investigators, and other researchers will remain blind to the allocation of the study drug and placebo.
  If serious adverse events occur to subjects during the study, the investigator must be informed of the treatment received by the subjects before appropriate treatment can be given. For safety reasons, the investigator may unblind the subjects urgently after obtaining the consent of the sponsor's medical monitor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JS005 150mg (recombinant humanized monoclonal antibody against IL-17A) (Experimental)
  Interventions: Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A)
- JS005 300mg (recombinant humanized monoclonal antibody against IL-17A) (Experimental)
  Interventions: Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A)
- Placebo (Placebo Comparator)
  Interventions: Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A)

INTERVENTIONS:
Biological: JS005 (recombinant humanized monoclonal antibody against IL-17A) — JS005/placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled Phase III clinical study to evaluate the efficacy and safety of JS005 in 702 adult patients with moderate-to-severe chronic plaque psoriasis

DETAILED DESCRIPTION:
The study consisted of four periods: screening period (up to 4 weeks), induction period (12 weeks), maintenance period (40 weeks) and follow-up period (8 weeks). This study planned to recruit 702 subjects, who were randomized into JS005 300mg group (234 subjects), JS005 150mg group (234 subjects) and placebo group (234 subjects) at a ratio of 1:1:1, and were stratified by whether they had previsouly received biologic treatments (continuous biologic treatment for ≥3 months at recommended doses or intolerance for safety reasons) and body weight (≥70 kg or < 70 kg).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily particpate in this clinical study and sign the informed consent form.
2. Male and female patients aged 18-75 years at the time of screening (both inclusive).
3. Fertile female subjects must be willing to use a highly effective contraceptive method during the study period and 20 weeks (expected 5 half-lives) after the last study drug administration and have a negative pregnancy test during the screening period and prior to randomization.

Exclusion Criteria:

1. Pregnant and lactating women.
2. A history of inflammatory bowel disease or other conditions with a high risk of perforation (e.g., severe gastrointestinal ulcers, etc.) or with other active autoimmune diseases (e.g., systemic lupus erythematosus, Sarcoidosis, etc.).
3. Have a type of psoriasis other than chronic plaque psoriasis (e.g., pustular, erythrodermic, and guttate psoriasis), drug-induced psoriasis, or have an active inflammatory skin disease other than psoriasis
4. Use of phototherapy, including but not limited to ultraviolet A phototherapy (with or without psoralens), ultraviolet B phototherapy, or excimer laser within 4 weeks prior to randomization. Subjects are unwilling to avoid excessive sunlight exposure within 4 weeks prior to randomization and during the study period;
5. A (current) history of systemic infection or serious infection requiring hospitalization and/or intravenous anti-infective therapy (e.g., antibiotics, antifungal agents, antiviral agents) within 12 weeks prior to randomization; a history of any active infection, other than common upper respiratory infections, within 2 weeks prior to randomization;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Change in PASI 90 | From week 0 to week 12
  The proportion of patients who achieved at least 90% improvement from baseline in psoriasis area and severity index (PASI 90) at week 12
Change in sPGA | From week 0 to week 12
  The proportion of patients who achieved a static physician Comprehensive Assessment (sPGA) score of 0 or 1 at week 12.

SECONDARY OUTCOMES:
Patients achieving PASI 75 at Week 12 | From week 0 to week 12
  The proportion of patients who achieved at least 75% improvement from baseline in psoriasis area and severity index (PASI 90) at week 12
Patients achieving PASI 100 at Week 12 | From week 0 to week 12
  The proportion of patients who achieved at least 100% improvement from baseline in psoriasis area and severity index (PASI 90) at week 12
Proportion of subjects with a sPGA score of 0 at week 12 | From week 0 to week 12
  The proportion of patients who achieved at least 0 at week 12
Proportion of subjects with a DLQI score of 0/1 at week 12 | From week 0 to week 12
  The proportion of patients who with a DLQI score at least 0/1 at week 12
Patients achieving PASI 75 at Week 52 | From week 0 to week 52
  Proportion of participants with a PASI score improvement of at least 75% (PASI 75) from baseline at week 52
Time to PASI 75/90 response | From week 0 to week 12
  Time to PASI 75/90 response within 12 weeks
Time to sPGA 0/1 response | From week 0 to week 12
  Time to sPGA 0/1 response within 12 weeks
Patients achieving PASI 90 at Week 52 | From week 0 to week 52
  Proportion of participants with a PASI score improvement of at least 90 (PASI 90) from baseline at week 52
Patients achieving PASI 100 at Week 52 | From week 0 to week 52
  Proportion of participants with a PASI score improvement of at least 100 from baseline (PASI 100) at week 52

CONTACTS AND LOCATIONS:
Locations (63):
- China (63):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Beijing, Beijing Municipality
  - Beijing LuHe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Nanyang city first People's Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Shiyan City People's Hospital, Shiyan, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Xiangya Third Hospital, Central South University, Changsha, Hunan
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - Jiangxi Dermatology Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Bethune First Hospital of Jilin University, Changchun, Jilin
  - Panjin Liao oil precious stone flower hospital, Panjin, Liaoning
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Shenyang Hospital of Integrated Chinese and Western Medicine, Shenyang, Liaoning
  - North East Central International Hospital Limited, Shenyang, Liaoning
  - Baotou Central Hospital, Baotou, Neimenggu
  - Inner Mongolia Baotou Steel Hospital, Baotou, Neimengu
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - Shandong Dermatology Hospital, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University City:Taiyuan, Taiyuan, Shanxi
  - Medicine School of Xi'an Jiaotong University, Xian, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University City:Xian, Xi’an, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang